CLINICAL TRIAL: NCT03978143
Title: A PHASE 1, OPEN LABEL, CROSSOVER STUDY TO EVALUATE PALATABILITY AND RELATIVE BIOAVAILABILITY OF TWO PEDIATRIC MICROSPHERE FORMULATIONS OF CRIZOTINIB IN HEALTHY PARTICIPANTS
Brief Title: Evaluate Taste and Relative Bioavailability of Two Microsphere Formulations of Crizotinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A8081069
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: Adult; Bioavailability; Crizotinib; Drug Interactions; Esomeprazole; Humans; Microsphere; Pharmacokinetics; Safety; Taste

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Other): Receive treatments in the following order from Periods 1-6: A, B, C, D, E, G
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Treatment E; Drug: Treatment G
- Sequence 2 (Other): Receive treatments in the following order from Periods 1-6: A, C, B, D, E, G
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Treatment E; Drug: Treatment G
- Sequence 3 (Other): Receive treatments in the following order from Periods 1-6: B, A, C, D, E, G
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Treatment E; Drug: Treatment G
- Sequence 4 (Other): Receive treatments in the following order from Periods 1-6: B, C, A, D, F, H
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Treatment F; Drug: Treatment H
- Sequence 5 (Other): Receive treatments in the following order from Periods 1-6: C, A, B, D, F, H
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Treatment F; Drug: Treatment H
- Sequence 6 (Other): Receive treatments in the following order from Periods 1-6: C, B, A, D, F, H
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Treatment F; Drug: Treatment H

INTERVENTIONS:
Drug: Treatment A — Single 250 mg crizotinib dose as coated microsphere 1 (cMS1) formulation will be administered on the morning of Day 1 after an overnight fast of at least 10 hours.
Drug: Treatment B — A single 250 mg crizotinib dose as coated microsphere 2 (cMS2) formulation will be administered on the morning of Day 1 after overnight fast of at least 10 hours.
Drug: Treatment C — A single 250 mg crizotinib dose as FC formulation will be administered on the morning of Day 1 after an overnight fast of at least 10 hours.
Drug: Treatment D — A single 250 mg crizotinib dose as OS will be administered on the morning of Day 1 after an overnight fast of at least 10 hours.
Drug: Treatment E — 250 mg crizotinib as cMS1 formulation will be administered with high-fat, high-calorie meal after an overnight fast of at least 10 hours.
  Arms: Sequence 1; Sequence 2; Sequence 3
Drug: Treatment F — 250 mg crizotinib as cMS2 will be administered with a high-fat, high-calorie meal after an overnight fast of at least 10 hours.
  Arms: Sequence 4; Sequence 5; Sequence 6
Drug: Treatment G — 40 mg esomeprazole will be administered
  1 hour prior to dinner on Day -5 through Day -1. A single 250 mg crizotinib dose as cMS1 formulation will be administered on the morning of Day 1 after an overnight fast of at least 10 hours.
  Arms: Sequence 1; Sequence 2; Sequence 3
Drug: Treatment H — 40 mg esomeprazole will be administered
  1 hour prior to dinner on Day -5 through Day -1. A single 250 mg crizotinib dose as cMS2 formulation will be administered on the morning of Day 1 after an overnight fast of at least 10 hours.
  Arms: Sequence 4; Sequence 5; Sequence 6

SUMMARY:
The primary purpose of the study is to estimate the relative bioavailability and palatability of 2 new crizotinib formulations to the commercially available crizotinib formulated capsule at a 250 mg dose administered under fasted conditions in adult healthy participants. Additionally, this study aims to assess the safety and tolerability of crizotinib 250 mg single dose in 4 formulations when given fasted, with high fat meal, or with a proton pump inhibitor in healthy participants. Finally, this study will explore the effect of food or proton pump inhibitor on the pharmacokinetics of the 2 new crizotinib formulations.

We hypothesize 1 of the 2 new crizotinib formulations will have improved relative bioavailability and palatability than the formulated capsule under fasted or fed conditions with or without a proton pump inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, gastric or intestinal bypass surgery, cholecystectomy).
* Any condition possibly affecting the ability to taste (eg, dysgeusia, respiratory infection).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory test abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of crizotinib.
* Participants with history of known sensitivity to esomeprazole or substituted benzimidazoles.
* Previous administration with an investigational product within 30 days or 5 half-lives preceding the first dose of crizotinib (whichever is longer).
* A positive urine drug test or cotinine test.
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Baseline 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QT interval corrected using the Fridericia's method [QTcF] >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If QTcF exceeds 450 msec, or the QRS complex exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS complex values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary: Aspartate aminotransferase (AST) or ALT level ≥1.5 × upper limit of normal (ULN); Total bilirubin (TBili) level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN; Estimated glomerular filtration rate (eGFR) <60 ml/min/1.73 m2 (See Appendix 10.2 for calculation method).
* Male participants who are unwilling or unable to comply with the contraception requirement listed in Section 10.4.1.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer,

  1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Participants who currently smoke.
* Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 0 (pre-dose), 1, 2, 4, 6, 8, 10, 12, 24, 48, and 96 hours post-dose in Periods 1, 2, 3, 5, and 6.
  AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0 (pre-dose), 1, 2, 4, 6, 8, 10, 12, 24, 48, and 96 hours post-dose in Periods 1, 2, 3, 5, and 6.
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Maximum Observed Plasma Concentration (Cmax) | 0 (pre-dose), 1, 2, 4, 6, 8, 10, 12, 24, 48, and 96 hours post-dose in Periods 1, 2, 3, 5, and 6.
  Maximum observed plasma concentration.
Number of subjects reporting overall liking of drug formulation | 1 (immediately after dosing), 5, 10, and 20 minutes after crizotinib administration in Treatments A, B and D.
  Overall liking assesses the degree that a participant likes a drug formulation based on sensory attributes experienced by the participant after tasting a product. It is scored based on a measurement of taste questionnaire.
Number of subjects reporting bitterness of drug formulation | 1 (immediately after dosing), 5, 10, and 20 minutes after crizotinib administration in Treatments A, B and D.
  Bitterness assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire.
Number of subjects reporting mouth feel from drug formulation | 1 (immediately after dosing), 5, 10, and 20 minutes after crizotinib administration in Treatments A, B and D.
  Mouth feel assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire.
Number of subjects reporting tongue/mouth burn from drug formulation | 1 (immediately after dosing), 5, 10, and 20 minutes after crizotinib administration in Treatments A, B and D.
  Tongue/mouth burn assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire.
Number of subjects reporting throat burn from drug formulation | 1 (immediately after dosing), 5, 10, and 20 minutes after crizotinib administration in Treatments A, B and D.
  Throat burn assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire.
Percentage of subjects reporting overall liking of drug formulation | 1 (immediately after dosing), 5, 10, and 20 minutes after crizotinib administration in Treatments A, B and D.
  Overall liking assesses the degree that a participant likes a drug formulation based on sensory attributes experienced by the participant after tasting a product. It is scored based on a measurement of taste questionnaire.
Percentage of subjects reporting bitterness of drug formulation | 1 (immediately after dosing), 5, 10, and 20 minutes after crizotinib administration in Treatments A, B and D.
  Bitterness assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire.
Percentage of subjects reporting mouth feel from drug formulation | 1 (immediately after dosing), 5, 10, and 20 minutes after crizotinib administration in Treatments A, B and D.
  Mouth feel assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire.
Percentage of subjects reporting tongue/mouth burn from drug formulation | 1 (immediately after dosing), 5, 10, and 20 minutes after crizotinib administration in Treatments A, B and D.
  Tongue/mouth burn assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire.
Percentage of subjects reporting throat burn from drug formulation | 1 (immediately after dosing), 5, 10, and 20 minutes after crizotinib administration in Treatments A, B and D.
  Throat burn assesses the degree that a participant experienced this sensory attribute after tasting a drug formulation. It is scored based on a measurement of taste questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A8081069